CLINICAL TRIAL: NCT05526209
Title: Longitudinal Relaxing Incision as a Technique for Recurrence Prevention in Ventral Hernia... Does it Help?
Brief Title: Longitudinal Relaxing Incision as a Technique for Recurrence Prevention in Ventral Hernia
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Mostafa Hussien Mohamed sabry Hussien, resident, Assiut University
Other Study IDs: Ventral Hernia
Record Dates: First submitted 2022-08-23; First posted 2022-09-02 (Actual); Last update posted 2022-09-02 (Actual); Status verified 2022-08

CONDITIONS: Ventral Hernia
MeSH Terms: conditions — Hernia, Ventral

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- 1 with using longitudinal relaxing incision: using longitudinal relaxing incision as a technique for recurrence prevention in ventral hernia
  Interventions: Procedure: using longitudinal relaxing incision as a technique for recurrence prevention in ventral hernia
- 2 without using longitudinal relaxing incision: without using longitudinal relaxing incision as a technique for recurrence prevention in ventral hernia

INTERVENTIONS:
Procedure: using longitudinal relaxing incision as a technique for recurrence prevention in ventral hernia — using longitudinal relaxing incision as a technique for recurrence prevention in ventral hernia
  Groups: 1 with using longitudinal relaxing incision

SUMMARY:
The aim of the study is showing the efficiency of using Longitudinal relaxing incision as a Technique for recurrence prevention in Ventral Hernia

DETAILED DESCRIPTION:
Ventral hernias of the abdomen are defined as a non-inguinal, nonhiatal defect in the fascia of the abdominal wall. Annually, there are about 350,000 ventral hernia operations. The repair of these abdominal wall defects is a common surgery performed by general surgeons. Surgery is typically recommended for individuals with acceptable operative risk, symptomatic hernias, or those at elevated risk of developing complications from a hernia. They can affect an individual's quality of life and can lead to hospitalizations and even death in some cases Etiologies of a ventral hernia can be broken down into 2 main categories; acquired or congenital. The vast majority of hernias that general surgeons see and treat are acquired; however, some individuals live with their ventral hernias from birth for prolonged periods of time before having them surgically repaired. Common causes of acquired ventral hernias include previous surgery causing an incisional hernia, trauma, and repetitive stress on naturally weak points of the abdominal wall. These naturally occurring weak points in the abdominal wall include the umbilicus, semilunar line, ostomy sites, bilateral inguinal regions, and esophageal hiatus. Obesity is a large component of hernias as well because it stretches the fascia of the abdomen causing it to weaken. Specifically, the action of repetitive weight gain and loss leads to weakening The most common treatment of ventral hernias includes surgery. Asymptomatic hernias are repaired on an elective basis, but those presenting with strangulation require immediate surgery. Incarceration without strangulation is not a surgical emergency; however, the risks and benefits of surgery should be discussed with the patient, and a patient with reasonable operative risk should have their hernia repaired within a sensible time frame. Non-surgical management of abdominal wall hernias with the use of binders, trusses, or corsets is not considered to be effective. However, this may be the only option in a patient who is not a reasonable candidate for surgery Over the years, many types of surgical techniques have been developed to repair hernias. There are many tenants of hernia repair. The most important being a tension-free closure, but others include the use of a mesh with 3 to 5 cm of overlap, meticulous handling of the mesh, preventing surgical site infections, and using a sublay technique with the closure of the fascia if possible. The most basic approach is a primary open repair without mesh, which should typically be reserved for defects in the fascia of less than 2 cm. An open repair with mesh has several options including what type of mesh and where to place the mesh.

Hernia recurrence is an extremely important postoperative outcome and assesses surgical efficacy. The ability to predict recurrence accurately would have considerable clinical utility, allowing surgeons to make better-informed decisions with their patients as to when and when not, to operate.

Multiple associated conditions, such as obesity, smoking, and others, have been reported in various studies to contribute to higher recurrence rates.

ELIGIBILITY:
Inclusion Criteria:

* any patient with Ventral Hernia admitted at Assiut University Hospital

Exclusion Criteria:

* recurrent hernia
* complicated [obstructed & strangulated]

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: cases with Ventral Hernia admitted at Assiut University Hospital at the period of the study
Sampling Method: Non-Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2022-09-01 (Estimated); Primary Completion 2023-12 (Estimated); Study Completion 2024-05 (Estimated)

PRIMARY OUTCOMES:
longitudinal relaxing incision | baseline
  the efficiency of using longitudinal relaxing incision as a technique for recurrence prevention in ventral hernia

REFERENCES:
- [Background] Cho JE, Helm MC, Helm JH, Mier N, Kastenmeier AS, Gould JC, Goldblatt MI. Retro-rectus placement of bio-absorbable mesh improves patient outcomes. Surg Endosc. 2019 Aug;33(8):2629-2634. doi: 10.1007/s00464-018-6560-y. Epub 2018 Oct 25. PMID 30361969
- [Background] Petro CC, Haskins IN, Perez AJ, Tastaldi L, Strong AT, Ilie RN, Tu C, Krpata DM, Prabhu AS, Eghtesad B, Rosen MJ. Hernia repair in patients with chronic liver disease - A 15-year single-center experience. Am J Surg. 2019 Jan;217(1):59-65. doi: 10.1016/j.amjsurg.2018.10.020. Epub 2018 Oct 16. PMID 30343877
- [Background] Schlosser KA, Arnold MR, Otero J, Prasad T, Lincourt A, Colavita PD, Kercher KW, Heniford BT, Augenstein VA. Deciding on Optimal Approach for Ventral Hernia Repair: Laparoscopic or Open. J Am Coll Surg. 2019 Jan;228(1):54-65. doi: 10.1016/j.jamcollsurg.2018.09.004. Epub 2018 Oct 22. PMID 30359827
- [Background] Berrevoet F. Prevention of Incisional Hernias after Open Abdomen Treatment. Front Surg. 2018 Feb 26;5:11. doi: 10.3389/fsurg.2018.00011. eCollection 2018. PMID 29536013
- [Background] Heniford BT. SAGES guidelines for laparoscopic ventral hernia repair. Surg Endosc. 2016 Aug;30(8):3161-2. doi: 10.1007/s00464-016-5073-9. Epub 2016 Jul 15. No abstract available. PMID 27422242
- [Background] Souza JM, Dumanian GA. Routine use of bioprosthetic mesh is not necessary: a retrospective review of 100 consecutive cases of intra-abdominal midweight polypropylene mesh for ventral hernia repair. Surgery. 2013 Mar;153(3):393-9. doi: 10.1016/j.surg.2012.08.003. Epub 2012 Oct 13. PMID 23068089
- [Background] de Vries HS, Smeeing D, Lourens H, Kruyt PM, Mollen RMHG. Long-term clinical experience with laparoscopic ventral hernia repair using a ParietexTM composite mesh in severely obese and non-severe obese patients: a single center cohort study. Minim Invasive Ther Allied Technol. 2019 Oct;28(5):304-308. doi: 10.1080/13645706.2018.1521431. Epub 2018 Oct 11. PMID 30307356
- [Background] Bencini L, Sanchez LJ, Bernini M, Miranda E, Farsi M, Boffi B, Moretti R. Predictors of recurrence after laparoscopic ventral hernia repair. Surg Laparosc Endosc Percutan Tech. 2009 Apr;19(2):128-32. doi: 10.1097/SLE.0b013e31819cb04b. PMID 19390279